CLINICAL TRIAL: NCT05169736
Title: Internet-based Cognitive Behavioural Therapy for Mental Health Problems Related to the Climate Crisis
Brief Title: ICBT for Mental Health Problems Related to the Climate Crisis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ClimateCope
Record Dates: First submitted 2021-12-20; First posted 2021-12-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Depression and Quality of Life
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based Cognitive Behavior Therapy (Experimental): ICBT, were participants receive 8 out of 15 possible modules, depending on their current problems and needs, 8 week long internet intervention for coping with mental health issues related to the climate crisis.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Wait-list control (No Intervention): Participants in the control group will be instructed to wait. Once intervention group will be finished, participants in control group will be able to access the same intervention.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Intervention based on cognitive behavioural therapy principles and adapted to mental health problems related to the climate crisis. Intervention's main purpose is to increase management of mental health issues such as depressive symtoms, stress, worry and anxiety related to the coronavirus pandemic and increase quality of life in the current situation. Intervention contains psycho-educational elements as well as examples and exercises.
  Arms: Internet-based Cognitive Behavior Therapy

SUMMARY:
The study seeks to investigate the effects of a guided internet-based cognitive behavioral therapy (ICBT) programme on adult mental health problems related to the climate crisis. ICBT will be compared to a wait-list control group.

Participants will be recruited in Sweden with a nationwide recruitment.

DETAILED DESCRIPTION:
The study is set up as a randomized controlled trial. Quality of life, depressive symptoms, anxiety, sleep problems and traumatic stress will be measured. Given uncertainties regarding the psychological effects connected to the climate crisis, a transproblematic tailored treatment approach will be used that has been tested in several previous trials. However, the present program has been adapted for the target population of people who are affected directly or indirectly by the societal and individual consequences of the climate crisis.

ELIGIBILITY:
Inclusion Criteria:

Experience mental health problems that are caused or exacerbated by the climate crisis and/or its consequences 18 years or older. Adequate ability to understand and speak Swedish. Access to the internet and a smartphone/computer.

Exclusion Criteria:

Other ongoing psychological treatment or counselling that interfere with trial treatment.

Recent (within the past 3 months) changes in the dose of psychotropic medication.

Any severe psychiatric or somatic conditions that would interfere with trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-06-27 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Becks Depression Inventory-II | Baseline, 8 weeks and follow-up at 12 months after treatment termination
  Measure of depressive symptoms. Possible range for the total sum: 0 to 63 (created by summing up the score from each item) with a higher score indicating a higher level of depressive symptoms. Clinical ranges for minimal, mild, moderate and severe major depressive disorder are considered to be 0-13, 13-19, 20-28, and 29-63 points.
Change in Perceived Stress Scale | Baseline, 8 weeks and follow-up at 12 months after treatment termination.
  It is a measure of the degree to which situations in one's life are appraised as stressful. It contains 10 items that are scored on a range between 0 (never) to 4 (very often). The total score can range from 0-56 and a higher score reflects higher levels of perceived stress.
Change in Generalised Anxiety Disorder 7-item scale | Baseline, 8 weeks and follow-up at 12 months after treatment termination.
  Seven item measure of generalized anxiety disorder. Sum score range from 0 to 21, with higher scores indicating more generalized anxiety. Cut-offs for interpretation: 0-5 minimal anxiety, 6-9 mild anxiety, 10-14 moderate anxiety, and 15-21 severe anxiety.

SECONDARY OUTCOMES:
Change in Insomnia Severity Index | Baseline, 8 weeks and follow-up at 12 months after treatment termination.
  Measure of insomnia severity and symptoms of disordered sleep. The total score can range between 0 (no sleep problems) to 28 (severe sleep problems and insomnia) with higher scores indicating severer levels of sleeping problems. Norm score ranges include low likelihood of sleep problems (0 to 7 points), some sleep problems (8 to 14 points), moderate sleep problems (15 to 21 points), severe sleep problems (22 to 28 points).
Change in Patient Health Questionnaire | Baseline, 8 weeks and follow-up at 12 months after treatment termination.
  Measure of depressive symptoms. Possible range for the total sum: 0 to 27 (created by summing up the score from each item) with a higher score indicating higher levels of depression. Clinical cut-offs for mild, moderate, moderately severe and severe major depressive disorder are considered to be 5, 10, 15, and 20 points.
Change in Alcohol Use Disorder Identification Test | Baseline, 8 weeks and follow-up at 12 months after treatment termination.
  The Alcohol Use Disorders Identification Test is a 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. 10 items and scores ranging from 0-40 with higher scores indicating a higher level of alcohol use.
Change in ClimateCope Index (CCI) | Baseline, 8 weeks and follow-up at 12 months after treatment termination
  This scale was constructed by the research group, measuring coping strategies connected to the climate situations. It is a 33 item scale rating from 1 (not at all) to 5 (totally agree), with higher scores indicating more helpful coping strategies.
Change in Brunnsviken Brief Quality of Life Scale | Baseline, 8 weeks and follow-up at 12 months after treatment termination
  Measure of quality of life, total score ranging from 0 to 96 with a higher score indicating a higher quality of life. The scores of each of the six primary questions regarding perceived quality of life within an area of life are multiplied with the score of an item measuring the perceived importance of the area in question.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Principal Investigator — Linkoeping University
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden